CLINICAL TRIAL: NCT00037765
Title: Gene Modifiers of Cystic Fibrosis Lung Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00-1420; 5R01HL068890 (NIH)
Record Dates: First submitted 2002-05-20; First posted 2002-05-21 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis; Lung Diseases
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine genetic modifiers of the severity of cystic fibrosis lung disease.

DETAILED DESCRIPTION:
BACKGROUND:

Cystic Fibrosis is caused by mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene resulting in impaired chloride transport across epithelial cells. While many organs are involved, infection, inflammation and destruction of the lungs ultimately result in morbidity and mortality. There is an association between residual CFTR function and severity of disease, however there is great variability within specific mutations suggesting gene modifiers. Even though there are over 900 mutations in CFTR that are related to CF lung disease, F508 the most common one is represented in 70 percent of the American CF population. Thus, establishing a phenotype/genotype correlation using homozygote F508 patients is likely to identify genes that are responsible for a mild form of disease. Why is this important? Whereas since the identification of the gene CFTR a significant amount of knowledge has been accumulated on CFTR function and CF pathogenesis, the cure for CF (treated as a monogenic disease) has been elusive. Identification of genetic modifiers (that may explain why 10 percent of CF patients died before the age of 10, 1/3 before the age of 20 while 50 percent live over 32 years of age) should expand the therapeutic targets that may lead to shifting of the severe phenotypes to milder ones. Moreover, the approach outlined in this study may also result in a better understanding of CFTR and delta F508 biogenesis and function, as it may identify genes directly related to CFTR.

The study is in response to a Request for Applications titled "Genetic Modifiers of Single Gene Defect Diseases" released in August, 2000 and co-sponsored by the National Institute of Diabetes, Digestive, and Kidney Diseases.

DESIGN NARRATIVE:

Patients with cystic fibrosis (CF) display a wide range of disease severity, particularly in pulmonary phenotype. Although some of this variability can be attributed to specific mutations within the CFTR gene (allelic heterogeneity), much of this variability has not been adequately explained. The central hypothesis of the study is that much of the "severity" (or "mildness") of CF lung disease reflects the influence of non-CFTR "modifier" alleles (genes). The study is designed to identify associations between non-CFTR genes and the pulmonary phenotype. To accomplish this goal, studies will be conducted on 600 CF patients who have the same CFTR genetic background, i.e., homozygous deltaF508, and who are at the extremes of pulmonary phenotype, i.e., the most severe and mildest lung disease. Pulmonary disease severity (or mildness) will be quantitated by longitudinal lung function analysis with informative censoring. The overall strategy will be to test for the association of candidate modifier alleles (genes) with the severity (or mildness) of pulmonary disease. Key clinical features (gender; age-at-diagnosis; sweat chloride; nutrition; and respiratory microbiology) will be important variables in the overall analysis. Initially, the study will test candidate genes (n=200) that have been implicated in the pathophysiology of CF lung disease. A pooling strategy will be used to expedite the first rounds of testing. After pooling DNA from the "severe" patients, and pooling DNA from the mild patients, those genes (alleles) can be identified with the greatest association with phenotype. Follow-up genotyping in individual subjects will allow subgroup analyses (gender; age-at-diagnosis; nutrition; respiratory microbiology) for each gene, as well as more complex analyses to search for interaction among different alleles. Subsequent studies will involve genome-wide testing with single nucleotide polymorphisms (SNPs) to identify loci (and genes) that are not present in the initial list of candidate genes. Identification of genes that modulate the severity of the pulmonary phenotype will improve understanding of the pathophysiology of CF lung disease, and identify new targets for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CF

Exclusion criteria:

* Only those subjects who are not able to consent to this protocol

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients who have the same CFTR genetic background, i.e., homozygous F508del, and who are at the extremes of pulmonary phenotype, i.e., the most severe and mildest lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2001-09; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
This is not an interventional study. | This is not an interventional study
  Not applicable. This is not an interventional study.

CONTACTS AND LOCATIONS:
Overall Officials: Wanda K O'Neal, PhD, Principal Investigator — University of North Carolina
Locations (1):
- Marsico Lung Institute, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Mencin A, Seki E, Osawa Y, Kodama Y, De Minicis S, Knowles M, Brenner DA. Alpha-1 antitrypsin Z protein (PiZ) increases hepatic fibrosis in a murine model of cholestasis. Hepatology. 2007 Nov;46(5):1443-52. doi: 10.1002/hep.21832. PMID 17668872
- [Background] Vecchio-Pagan B, Blackman SM, Lee M, Atalar M, Pellicore MJ, Pace RG, Franca AL, Raraigh KS, Sharma N, Knowles MR, Cutting GR. Deep resequencing of CFTR in 762 F508del homozygotes reveals clusters of non-coding variants associated with cystic fibrosis disease traits. Hum Genome Var. 2016 Nov 24;3:16038. doi: 10.1038/hgv.2016.38. eCollection 2016. PMID 27917292
- [Background] Collaco JM, Raraigh KS, Appel LJ, Cutting GR. Respiratory pathogens mediate the association between lung function and temperature in cystic fibrosis. J Cyst Fibros. 2016 Nov;15(6):794-801. doi: 10.1016/j.jcf.2016.05.012. Epub 2016 Jun 11. PMID 27296562
- [Background] Gong J, Wang F, Xiao B, Panjwani N, Lin F, Keenan K, Avolio J, Esmaeili M, Zhang L, He G, Soave D, Mastromatteo S, Baskurt Z, Kim S, O'Neal WK, Polineni D, Blackman SM, Corvol H, Cutting GR, Drumm M, Knowles MR, Rommens JM, Sun L, Strug LJ. Genetic association and transcriptome integration identify contributing genes and tissues at cystic fibrosis modifier loci. PLoS Genet. 2019 Feb 26;15(2):e1008007. doi: 10.1371/journal.pgen.1008007. eCollection 2019 Feb. PMID 30807572
- [Background] Darrah RJ, Jacono FJ, Joshi N, Mitchell AL, Sattar A, Campanaro CK, Litman P, Frey J, Nethery DE, Barbato ES, Hodges CA, Corvol H, Cutting GR, Knowles MR, Strug LJ, Drumm ML. AGTR2 absence or antagonism prevents cystic fibrosis pulmonary manifestations. J Cyst Fibros. 2019 Jan;18(1):127-134. doi: 10.1016/j.jcf.2018.05.013. Epub 2018 Jun 22. PMID 29937318
- [Background] Panjwani N, Xiao B, Xu L, Gong J, Keenan K, Lin F, He G, Baskurt Z, Kim S, Zhang L, Esmaeili M, Blackman S, Scherer SW, Corvol H, Drumm M, Knowles M, Cutting G, Rommens JM, Sun L, Strug LJ. Improving imputation in disease-relevant regions: lessons from cystic fibrosis. NPJ Genom Med. 2018 Mar 20;3:8. doi: 10.1038/s41525-018-0047-6. eCollection 2018. PMID 29581887
- [Result] Drumm ML, Konstan MW, Schluchter MD, Handler A, Pace R, Zou F, Zariwala M, Fargo D, Xu A, Dunn JM, Darrah RJ, Dorfman R, Sandford AJ, Corey M, Zielenski J, Durie P, Goddard K, Yankaskas JR, Wright FA, Knowles MR; Gene Modifier Study Group. Genetic modifiers of lung disease in cystic fibrosis. N Engl J Med. 2005 Oct 6;353(14):1443-53. doi: 10.1056/NEJMoa051469. PMID 16207846
- [Result] Taylor-Cousar JL, Zariwala MA, Burch LH, Pace RG, Drumm ML, Calloway H, Fan H, Weston BW, Wright FA, Knowles MR; Gene Modifier Study Group. Histo-blood group gene polymorphisms as potential genetic modifiers of infection and cystic fibrosis lung disease severity. PLoS One. 2009;4(1):e4270. doi: 10.1371/journal.pone.0004270. Epub 2009 Jan 26. PMID 19169360
- [Result] Levy H, Murphy A, Zou F, Gerard C, Klanderman B, Schuemann B, Lazarus R, Garcia KC, Celedon JC, Drumm M, Dahmer M, Quasney M, Schneck K, Reske M, Knowles MR, Pier GB, Lange C, Weiss ST. IL1B polymorphisms modulate cystic fibrosis lung disease. Pediatr Pulmonol. 2009 Jun;44(6):580-93. doi: 10.1002/ppul.21026. PMID 19431193
- [Result] Gu Y, Harley IT, Henderson LB, Aronow BJ, Vietor I, Huber LA, Harley JB, Kilpatrick JR, Langefeld CD, Williams AH, Jegga AG, Chen J, Wills-Karp M, Arshad SH, Ewart SL, Thio CL, Flick LM, Filippi MD, Grimes HL, Drumm ML, Cutting GR, Knowles MR, Karp CL. Identification of IFRD1 as a modifier gene for cystic fibrosis lung disease. Nature. 2009 Apr 23;458(7241):1039-42. doi: 10.1038/nature07811. Epub 2009 Feb 25. PMID 19242412
- [Result] Li W, Sun L, Corey M, Zou F, Lee S, Cojocaru AL, Taylor C, Blackman SM, Stephenson A, Sandford AJ, Dorfman R, Drumm ML, Cutting GR, Knowles MR, Durie P, Wright FA, Strug LJ. Understanding the population structure of North American patients with cystic fibrosis. Clin Genet. 2011 Feb;79(2):136-46. doi: 10.1111/j.1399-0004.2010.01502.x. PMID 20681990
- [Result] Wright FA, Strug LJ, Doshi VK, Commander CW, Blackman SM, Sun L, Berthiaume Y, Cutler D, Cojocaru A, Collaco JM, Corey M, Dorfman R, Goddard K, Green D, Kent JW Jr, Lange EM, Lee S, Li W, Luo J, Mayhew GM, Naughton KM, Pace RG, Pare P, Rommens JM, Sandford A, Stonebraker JR, Sun W, Taylor C, Vanscoy LL, Zou F, Blangero J, Zielenski J, O'Neal WK, Drumm ML, Durie PR, Knowles MR, Cutting GR. Genome-wide association and linkage identify modifier loci of lung disease severity in cystic fibrosis at 11p13 and 20q13.2. Nat Genet. 2011 Jun;43(6):539-46. doi: 10.1038/ng.838. Epub 2011 May 22. PMID 21602797
- [Result] Schluchter MD, Konstan MW, Drumm ML, Yankaskas JR, Knowles MR. Classifying severity of cystic fibrosis lung disease using longitudinal pulmonary function data. Am J Respir Crit Care Med. 2006 Oct 1;174(7):780-6. doi: 10.1164/rccm.200512-1919OC. Epub 2006 Jul 20. PMID 16858011
- [Result] Knowles MR. Gene modifiers of lung disease. Curr Opin Pulm Med. 2006 Nov;12(6):416-21. doi: 10.1097/01.mcp.0000245707.59138.40. PMID 17053491
- [Result] Bartling TR, Drumm ML. Oxidative stress causes IL8 promoter hyperacetylation in cystic fibrosis airway cell models. Am J Respir Cell Mol Biol. 2009 Jan;40(1):58-65. doi: 10.1165/rcmb.2007-0464OC. Epub 2008 Jul 17. PMID 18635816
- [Result] Hillian AD, Londono D, Dunn JM, Goddard KA, Pace RG, Knowles MR, Drumm ML; CF Gene Modifier Study Group. Modulation of cystic fibrosis lung disease by variants in interleukin-8. Genes Immun. 2008 Sep;9(6):501-8. doi: 10.1038/gene.2008.42. Epub 2008 Jun 19. PMID 18563170
- [Result] Darrah R, McKone E, O'Connor C, Rodgers C, Genatossio A, McNamara S, Gibson R, Stuart Elborn J, Ennis M, Gallagher CG, Kalsheker N, Aitken M, Wiese D, Dunn J, Smith P, Pace R, Londono D, Goddard KA, Knowles MR, Drumm ML. EDNRA variants associate with smooth muscle mRNA levels, cell proliferation rates, and cystic fibrosis pulmonary disease severity. Physiol Genomics. 2010 Mar 3;41(1):71-7. doi: 10.1152/physiolgenomics.00185.2009. Epub 2009 Dec 22. PMID 20028935
- [Result] Bezzerri V, d'Adamo P, Rimessi A, Lanzara C, Crovella S, Nicolis E, Tamanini A, Athanasakis E, Tebon M, Bisoffi G, Drumm ML, Knowles MR, Pinton P, Gasparini P, Berton G, Cabrini G. Phospholipase C-beta3 is a key modulator of IL-8 expression in cystic fibrosis bronchial epithelial cells. J Immunol. 2011 Apr 15;186(8):4946-58. doi: 10.4049/jimmunol.1003535. Epub 2011 Mar 16. PMID 21411730
- [Result] Harris WT, Muhlebach MS, Oster RA, Knowles MR, Clancy JP, Noah TL. Plasma TGF-beta(1) in pediatric cystic fibrosis: potential biomarker of lung disease and response to therapy. Pediatr Pulmonol. 2011 Jul;46(7):688-95. doi: 10.1002/ppul.21430. Epub 2011 Feb 18. PMID 21337732
- [Result] Harris WT, Muhlebach MS, Oster RA, Knowles MR, Noah TL. Transforming growth factor-beta(1) in bronchoalveolar lavage fluid from children with cystic fibrosis. Pediatr Pulmonol. 2009 Nov;44(11):1057-64. doi: 10.1002/ppul.21079. PMID 19830844
- [Result] Guo X, Pace RG, Stonebraker JR, Commander CW, Dang AT, Drumm ML, Harris A, Zou F, Swallow DM, Wright FA, O'Neal WK, Knowles MR. Mucin variable number tandem repeat polymorphisms and severity of cystic fibrosis lung disease: significant association with MUC5AC. PLoS One. 2011;6(10):e25452. doi: 10.1371/journal.pone.0025452. Epub 2011 Oct 6. PMID 21998660
- [Result] Bartlett JR, Friedman KJ, Ling SC, Pace RG, Bell SC, Bourke B, Castaldo G, Castellani C, Cipolli M, Colombo C, Colombo JL, Debray D, Fernandez A, Lacaille F, Macek M Jr, Rowland M, Salvatore F, Taylor CJ, Wainwright C, Wilschanski M, Zemkova D, Hannah WB, Phillips MJ, Corey M, Zielenski J, Dorfman R, Wang Y, Zou F, Silverman LM, Drumm ML, Wright FA, Lange EM, Durie PR, Knowles MR; Gene Modifier Study Group. Genetic modifiers of liver disease in cystic fibrosis. JAMA. 2009 Sep 9;302(10):1076-83. doi: 10.1001/jama.2009.1295. PMID 19738092
- [Result] Blackman SM, Hsu S, Ritter SE, Naughton KM, Wright FA, Drumm ML, Knowles MR, Cutting GR. A susceptibility gene for type 2 diabetes confers substantial risk for diabetes complicating cystic fibrosis. Diabetologia. 2009 Sep;52(9):1858-65. doi: 10.1007/s00125-009-1436-2. Epub 2009 Jul 8. PMID 19585101
- [Result] Taylor C, Commander CW, Collaco JM, Strug LJ, Li W, Wright FA, Webel AD, Pace RG, Stonebraker JR, Naughton K, Dorfman R, Sandford A, Blackman SM, Berthiaume Y, Pare P, Drumm ML, Zielenski J, Durie P, Cutting GR, Knowles MR, Corey M. A novel lung disease phenotype adjusted for mortality attrition for cystic fibrosis genetic modifier studies. Pediatr Pulmonol. 2011 Sep;46(9):857-69. doi: 10.1002/ppul.21456. Epub 2011 Apr 1. PMID 21462361
- [Result] Zou F, Lee S, Knowles MR, Wright FA. Quantification of population structure using correlated SNPs by shrinkage principal components. Hum Hered. 2010;70(1):9-22. doi: 10.1159/000288706. Epub 2010 Apr 23. PMID 20413978
- [Result] Corvol H, Blackman SM, Boelle PY, Gallins PJ, Pace RG, Stonebraker JR, Accurso FJ, Clement A, Collaco JM, Dang H, Dang AT, Franca A, Gong J, Guillot L, Keenan K, Li W, Lin F, Patrone MV, Raraigh KS, Sun L, Zhou YH, O'Neal WK, Sontag MK, Levy H, Durie PR, Rommens JM, Drumm ML, Wright FA, Strug LJ, Cutting GR, Knowles MR. Genome-wide association meta-analysis identifies five modifier loci of lung disease severity in cystic fibrosis. Nat Commun. 2015 Sep 29;6:8382. doi: 10.1038/ncomms9382. PMID 26417704
- [Result] Dang H, Gallins PJ, Pace RG, Guo XL, Stonebraker JR, Corvol H, Cutting GR, Drumm ML, Strug LJ, Knowles MR, O'Neal WK. Novel variation at chr11p13 associated with cystic fibrosis lung disease severity. Hum Genome Var. 2016 Jul 7;3:16020. doi: 10.1038/hgv.2016.20. eCollection 2016. PMID 27408752
- [Result] O'Neal WK, Gallins P, Pace RG, Dang H, Wolf WE, Jones LC, Guo X, Zhou YH, Madar V, Huang J, Liang L, Moffatt MF, Cutting GR, Drumm ML, Rommens JM, Strug LJ, Sun W, Stonebraker JR, Wright FA, Knowles MR. Gene expression in transformed lymphocytes reveals variation in endomembrane and HLA pathways modifying cystic fibrosis pulmonary phenotypes. Am J Hum Genet. 2015 Feb 5;96(2):318-28. doi: 10.1016/j.ajhg.2014.12.022. Epub 2015 Jan 29. PMID 25640674
- [Result] Guo X, Pace RG, Stonebraker JR, O'Neal WK, Knowles MR. Meconium ileus in cystic fibrosis is not linked to central repetitive region length variation in MUC1, MUC2, and MUC5AC. J Cyst Fibros. 2014 Dec;13(6):613-6. doi: 10.1016/j.jcf.2014.05.005. Epub 2014 Jun 8. PMID 24920497
- [Result] Blackman SM, Commander CW, Watson C, Arcara KM, Strug LJ, Stonebraker JR, Wright FA, Rommens JM, Sun L, Pace RG, Norris SA, Durie PR, Drumm ML, Knowles MR, Cutting GR. Genetic modifiers of cystic fibrosis-related diabetes. Diabetes. 2013 Oct;62(10):3627-35. doi: 10.2337/db13-0510. Epub 2013 May 13. PMID 23670970
- [Result] Sun L, Rommens JM, Corvol H, Li W, Li X, Chiang TA, Lin F, Dorfman R, Busson PF, Parekh RV, Zelenika D, Blackman SM, Corey M, Doshi VK, Henderson L, Naughton KM, O'Neal WK, Pace RG, Stonebraker JR, Wood SD, Wright FA, Zielenski J, Clement A, Drumm ML, Boelle PY, Cutting GR, Knowles MR, Durie PR, Strug LJ. Multiple apical plasma membrane constituents are associated with susceptibility to meconium ileus in individuals with cystic fibrosis. Nat Genet. 2012 May;44(5):562-9. doi: 10.1038/ng.2221. PMID 22466613
- [Result] Miller MR, Soave D, Li W, Gong J, Pace RG, Boelle PY, Cutting GR, Drumm ML, Knowles MR, Sun L, Rommens JM, Accurso F, Durie PR, Corvol H, Levy H, Sontag MK, Strug LJ. Variants in Solute Carrier SLC26A9 Modify Prenatal Exocrine Pancreatic Damage in Cystic Fibrosis. J Pediatr. 2015 May;166(5):1152-1157.e6. doi: 10.1016/j.jpeds.2015.01.044. Epub 2015 Mar 11. PMID 25771386
- [Result] Knowles MR, Drumm M. The influence of genetics on cystic fibrosis phenotypes. Cold Spring Harb Perspect Med. 2012 Dec 1;2(12):a009548. doi: 10.1101/cshperspect.a009548. PMID 23209180
- [Result] Emond MJ, Louie T, Emerson J, Chong JX, Mathias RA, Knowles MR, Rieder MJ, Tabor HK, Nickerson DA, Barnes KC; NHLBI GO Exome Sequencing Project; Go L, Gibson RL, Bamshad MJ. Exome Sequencing of Phenotypic Extremes Identifies CAV2 and TMC6 as Interacting Modifiers of Chronic Pseudomonas aeruginosa Infection in Cystic Fibrosis. PLoS Genet. 2015 Jun 5;11(6):e1005273. doi: 10.1371/journal.pgen.1005273. eCollection 2015 Jun. PMID 26047157
- [Result] Henderson LB, Doshi VK, Blackman SM, Naughton KM, Pace RG, Moskovitz J, Knowles MR, Durie PR, Drumm ML, Cutting GR. Variation in MSRA modifies risk of neonatal intestinal obstruction in cystic fibrosis. PLoS Genet. 2012;8(3):e1002580. doi: 10.1371/journal.pgen.1002580. Epub 2012 Mar 15. PMID 22438829
- [Result] Kingston H, Stilp AM, Gordon W, Broome J, Gogarten SM, Ling H, Barnard J, Dugan-Perez S, Ellinor PT, Gabriel S, Germer S, Gibbs RA, Gupta N, Rice K, Smith AV, Zody MC; Cystic Fibrosis Genome Project; NHLBI Trans-Omics for Precision Medicine (TOPMed) Consortium; Blackman SM, Cutting G, Knowles MR, Zhou YH, Rosenfeld M, Gibson RL, Bamshad M, Fohner A, Blue EE. Accounting for population structure in genetic studies of cystic fibrosis. HGG Adv. 2022 May 12;3(3):100117. doi: 10.1016/j.xhgg.2022.100117. eCollection 2022 Jul 14. PMID 35647563
- [Result] Sun Q, Liu W, Rosen JD, Huang L, Pace RG, Dang H, Gallins PJ, Blue EE, Ling H, Corvol H, Strug LJ, Bamshad MJ, Gibson RL, Pugh EW, Blackman SM, Cutting GR, O'Neal WK, Zhou YH, Wright FA, Knowles MR, Wen J, Li Y; Cystic Fibrosis Genome Project. Leveraging TOPMed imputation server and constructing a cohort-specific imputation reference panel to enhance genotype imputation among cystic fibrosis patients. HGG Adv. 2022 Jan 11;3(2):100090. doi: 10.1016/j.xhgg.2022.100090. eCollection 2022 Apr 14. PMID 35128485
- [Result] Raraigh KS, Aksit MA, Hetrick K, Pace RG, Ling H, O'Neal W, Blue E, Zhou YH, Bamshad MJ, Blackman SM, Gibson RL, Knowles MR, Cutting GR. Complete CFTR gene sequencing in 5,058 individuals with cystic fibrosis informs variant-specific treatment. J Cyst Fibros. 2022 May;21(3):463-470. doi: 10.1016/j.jcf.2021.10.011. Epub 2021 Nov 12. PMID 34782259
- [Result] Rosenfeld M, Faino AV, Onchiri F, Aksit MA, Blackman SM, Blue EE, Collaco JM, Gordon WW, Pace RG, Raraigh KS, Zhou YH, Cutting GR, Knowles MR, Bamshad MJ, Gibson RL. Comparing encounter-based and annualized chronic pseudomonas infection definitions in cystic fibrosis. J Cyst Fibros. 2022 Jan;21(1):40-44. doi: 10.1016/j.jcf.2021.07.020. Epub 2021 Aug 13. PMID 34393091
- [Result] Pandey JP, Namboodiri AM, Nietert PJ, Knowles MR, Pace RG, Pier GB. Immunoglobulin GM and KM allotypes are associated with antibody responses to Pseudomonas aeruginosa antigens in chronically infected cystic fibrosis patients. J Cyst Fibros. 2021 Nov;20(6):1080-1084. doi: 10.1016/j.jcf.2021.06.011. Epub 2021 Jul 7. PMID 34246573
- [Result] Eastman AC, Pace RG, Dang H, Aksit MA, Vecchio-Pagan B, Lam AN, O'Neal WK, Blackman SM, Knowles MR, Cutting GR. SLC26A9 SNP rs7512462 is not associated with lung disease severity or lung function response to ivacaftor in cystic fibrosis patients with G551D-CFTR. J Cyst Fibros. 2021 Sep;20(5):851-856. doi: 10.1016/j.jcf.2021.02.007. Epub 2021 Mar 2. PMID 33674211
- [Result] Dang H, Polineni D, Pace RG, Stonebraker JR, Corvol H, Cutting GR, Drumm ML, Strug LJ, O'Neal WK, Knowles MR. Mining GWAS and eQTL data for CF lung disease modifiers by gene expression imputation. PLoS One. 2020 Nov 30;15(11):e0239189. doi: 10.1371/journal.pone.0239189. eCollection 2020. PMID 33253230
- [Result] Aksit MA, Pace RG, Vecchio-Pagan B, Ling H, Rommens JM, Boelle PY, Guillot L, Raraigh KS, Pugh E, Zhang P, Strug LJ, Drumm ML, Knowles MR, Cutting GR, Corvol H, Blackman SM. Genetic Modifiers of Cystic Fibrosis-Related Diabetes Have Extensive Overlap With Type 2 Diabetes and Related Traits. J Clin Endocrinol Metab. 2020 May 1;105(5):1401-15. doi: 10.1210/clinem/dgz102. PMID 31697830
- [Result] Polineni D, Piccorelli AV, Hannah WB, Dalrymple SN, Pace RG, Durie PR, Ling SC, Knowles MR, Stonebraker JR. Analysis of a large cohort of cystic fibrosis patients with severe liver disease indicates lung function decline does not significantly differ from that of the general cystic fibrosis population. PLoS One. 2018 Oct 11;13(10):e0205257. doi: 10.1371/journal.pone.0205257. eCollection 2018. PMID 30307979
- [Result] Polineni D, Dang H, Gallins PJ, Jones LC, Pace RG, Stonebraker JR, Commander LA, Krenicky JE, Zhou YH, Corvol H, Cutting GR, Drumm ML, Strug LJ, Boyle MP, Durie PR, Chmiel JF, Zou F, Wright FA, O'Neal WK, Knowles MR. Airway Mucosal Host Defense Is Key to Genomic Regulation of Cystic Fibrosis Lung Disease Severity. Am J Respir Crit Care Med. 2018 Jan 1;197(1):79-93. doi: 10.1164/rccm.201701-0134OC. PMID 28853905
- [Result] Collaco JM, Blackman SM, Raraigh KS, Corvol H, Rommens JM, Pace RG, Boelle PY, McGready J, Sosnay PR, Strug LJ, Knowles MR, Cutting GR. Sources of Variation in Sweat Chloride Measurements in Cystic Fibrosis. Am J Respir Crit Care Med. 2016 Dec 1;194(11):1375-1382. doi: 10.1164/rccm.201603-0459OC. PMID 27258095
- [Result] Guo X, Zheng S, Dang H, Pace RG, Stonebraker JR, Jones CD, Boellmann F, Yuan G, Haridass P, Fedrigo O, Corcoran DL, Seibold MA, Ranade SS, Knowles MR, O'Neal WK, Voynow JA. Genome reference and sequence variation in the large repetitive central exon of human MUC5AC. Am J Respir Cell Mol Biol. 2014 Jan;50(1):223-32. doi: 10.1165/rcmb.2013-0235OC. PMID 24010879
- [Result] Emond MJ, Louie T, Emerson J, Zhao W, Mathias RA, Knowles MR, Wright FA, Rieder MJ, Tabor HK, Nickerson DA, Barnes KC; National Heart, Lung, and Blood Institute (NHLBI) GO Exome Sequencing Project; Lung GO; Gibson RL, Bamshad MJ. Exome sequencing of extreme phenotypes identifies DCTN4 as a modifier of chronic Pseudomonas aeruginosa infection in cystic fibrosis. Nat Genet. 2012 Jul 8;44(8):886-9. doi: 10.1038/ng.2344. PMID 22772370
- [Result] Zhou YH, Gallins PJ, Pace RG, Dang H, Aksit MA, Blue EE, Buckingham KJ, Collaco JM, Faino AV, Gordon WW, Hetrick KN, Ling H, Liu W, Onchiri FM, Pagel K, Pugh EW, Raraigh KS, Rosenfeld M, Sun Q, Wen J, Li Y, Corvol H, Strug LJ, Bamshad MJ, Blackman SM, Cutting GR, Gibson RL, O'Neal WK, Wright FA, Knowles MR. Genetic Modifiers of Cystic Fibrosis Lung Disease Severity: Whole-Genome Analysis of 7,840 Patients. Am J Respir Crit Care Med. 2023 May 15;207(10):1324-1333. doi: 10.1164/rccm.202209-1653OC. PMID 36921087
- [Result] Sun Q, Yang Y, Rosen JD, Jiang MZ, Chen J, Liu W, Wen J, Raffield LM, Pace RG, Zhou YH, Wright FA, Blackman SM, Bamshad MJ, Gibson RL, Cutting GR, Knowles MR, Schrider DR, Fuchsberger C, Li Y. MagicalRsq: Machine-learning-based genotype imputation quality calibration. Am J Hum Genet. 2022 Nov 3;109(11):1986-1997. doi: 10.1016/j.ajhg.2022.09.009. Epub 2022 Oct 4. PMID 36198314
- [Result] Aksit MA, Ling H, Pace RG, Raraigh KS, Onchiri F, Faino AV, Pagel K, Pugh E, Stilp AM, Sun Q, Blue EE, Wright FA, Zhou YH, Bamshad MJ, Gibson RL, Knowles MR, Cutting GR, Blackman SM; CF Genome Project. Pleiotropic modifiers of age-related diabetes and neonatal intestinal obstruction in cystic fibrosis. Am J Hum Genet. 2022 Oct 6;109(10):1894-1908. doi: 10.1016/j.ajhg.2022.09.004. PMID 36206743